CLINICAL TRIAL: NCT04551105
Title: Evaluation of TaiHao Breast Ultrasound Diagnosis Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TaiHao Medical Inc. (Industry)
Collaborators: Columbia University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TaiHao BR-USCAD VT 20-249
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- First session: manual review first and then review with CADx (Active Comparator): Reader Group X interpret the "Dataset A" cases in different random order without any assistance of AI first, and then interpret the "Dataset B" cases in different random order with TaiHao AI system.
  Interventions: Diagnostic Test: Reader Group X - Session 1
- First session: review with CADx first and then manual review (Active Comparator): Reader Group Y interpret the "Dataset A" cases in different random order with TaiHao AI system first, and then interpret the "Dataset B" cases in different random order without any assistance of AI.
  Interventions: Diagnostic Test: Reader Group Y - Session 1
- Second session: manual review first and then review with CADx (Active Comparator): At least 4 weeks after first session for memory washing out. Reader Group X interpret the "Dataset A" cases in different random order with TaiHao AI system first, and then interpret the "Dataset B" cases in different random order without any assistance of AI.
  Interventions: Diagnostic Test: Reader Group X - Session 2
- Second session: review with CADx first and then manual review (Active Comparator): At least 4 weeks after first session for memory washing out. Rader Group Y interpret the "Dataset A" cases in different random order without any assistance of AI first, and then interpret the "Dataset B" cases in different random order with TaiHao AI system.
  Interventions: Diagnostic Test: Reader Group Y - Session 2

INTERVENTIONS:
Diagnostic Test: Reader Group X - Session 1 — Each rater in "Reader Group X" will interpret the "dataset A" cases in different random order without BR-USCAD DS and interpret the "dataset B" cases in different random order with BR-USCAD DS.
  Arms: First session: manual review first and then review with CADx
Diagnostic Test: Reader Group Y - Session 1 — Each rater in "Reader Group Y" will interpret the "dataset A" cases in different random order with BR-USCAD DS and interpret the "dataset B" cases in different random order without BR-USCAD DS.
  Arms: First session: review with CADx first and then manual review
Diagnostic Test: Reader Group X - Session 2 — Each rater in "Reader Group X" will interpret the "dataset A" cases in different random order with BR-USCAD DS and interpret the "dataset B" cases in different random order without BR-USCAD DS.
  Arms: Second session: manual review first and then review with CADx
Diagnostic Test: Reader Group Y - Session 2 — Each rater in "Reader Group Y" will interpret the "dataset A" cases in different random order without BR-USCAD DS and interpret the "dataset B" cases in different random order with BR-USCAD DS.
  Arms: Second session: review with CADx first and then manual review

SUMMARY:
The BR-USCAD DS Module is a computer-assisted detection and diagnosis software based on a deep learning algorithm. This retrospective, fully-crossed, multi-reader, multi-case (MRMC) study aims to compare the performances of readers without and with the aid of the Breast Ultrasound Image Reviewed with Assistance of Computer-Assisted Detection and Diagnosis System (BR-USCAD DS) in interpreting breast ultrasound images of lesions.

ELIGIBILITY:
Inclusion Criteria:

* B-mode breast ultrasound image
* Female, age 21 or older
* Breast lesion images acquired before a biopsy or surgery - these images were retrospectively collected with histology report.
* Non-biopsied benign lesions with negative follow-up for a minimum of 24 months
* At least two orthogonal views of a lesion

Exclusion Criteria:

* Breast lesion images acquired after biopsy or surgery.
* Any breast surgeries or interventional procedures in the 12 months prior to ultrasound imaging
* Case demonstrating administrative or technical errors
* Multiple lesions in one 2-D ultrasound image
* Breast ultrasound images with Doppler, elastography, or other overlays present
* Case with less than 2-year follow-up and without biopsy confirmation

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih Chung Lo, Ph.D., Study Director — Arlington Innovation Center: Health Research - Virginia Tech
Locations (1):
- Arlington Innovation Center: Health Research - Virginia Tech, Arlington, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six hundred and twenty-eight cases were randomized and split into two groups (A and B) with the same number of cases (314) in each group. Sixteen readers were randomized and split into two groups (X and Y) with the same number of readers (8) in each group.
Pre-assignment Details: 628 cases were randomly split into study datasets A and B. Each dataset had 314 cases. For each session, sub-datasets A and B were randomized within the group. Then, a reader read each sub-dataset either unaided or aided by the BU-CAD system.
Units Other Than Participants: cases
Groups:
- Arm 1: Group X readers read group A cases first unaided and then group B cases aided. At least 5 weeks later, group X readers read group B cases unaided, then group A cases aided.
- Arm2: Group Y readers read group B cases first unaided and then group A cases aided. At least 5 weeks later, group Y readers read group A cases unaided, then group B cases aided.
Period: The 1st Study Sessions
Arm/Group | Arm 1 | Arm2
Started | 8; 314 cases (Each reader of the same groups(8) tudy with the same number of cases (314).) | 8; 314 cases (Each reader of the same groups(8) tudy with the same number of cases (314).)
Completed | 8; 314 cases | 8; 314 cases
Not Completed | 0; 0 cases | 0; 0 cases
Period: The 2st Study Sessions (5 Weeks Later)
Arm/Group | Arm 1 | Arm2
Started | 8; 314 cases (Each reader of the same groups(8) tudy with the same number of cases (314).) | 8; 314 cases (Each reader of the same groups(8) tudy with the same number of cases (314).)
Completed | 8; 314 cases | 8; 314 cases
Not Completed | 0; 0 cases | 0; 0 cases

BASELINE CHARACTERISTICS:
Groups:
- Without BU-CAD Decision Support Assistance: Group X readers read group A cases(314) first unaided and then group B cases(314) aided. At least 5 weeks later, group X readers read group B cases(314) unaided, then group A cases(314) aided.
- With BU-CAD Decision Support Assistance: Group Y readers read group B cases(314) first unaided and then group A cases(314) aided. At least 5 weeks later, group Y readers read group A cases(314) unaided, then group B(314) cases aided.
- Total: Total of all reporting groups
Arm/Group | Without BU-CAD Decision Support Assistance | With BU-CAD Decision Support Assistance | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Area Under the LROC Curve
Description: The area under the LROC curve (AUC_LROC) on the diagnosis of benign and malignant lesions was computed and compared for Aim 1 (baseline) and Arm 2 (with BU-CAD assistance) studies.
Time Frame: 10 weeks
Population: Of the study breast ultrasound cases, some contained malignant lesions and some contained breast contained benign lesions.
Measure: Mean (95% Confidence Interval); unit: probability
Units Other Than Participants: case
Groups:
- Arm 1: read each breast ultrasound case without the BU-CAD decision support assistance referred to as the unaided (or baseline) study
- Arm 2: read each breast ultrasound case with the aid of BU-CAD decision support referred to as 'aided study
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 16
Number analyzed (case) | 628 | 628
probability | 0.7786 [0.7463 to 0.8109] | 0.8160 [0.7862 to 0.8458]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, OR-DBM model; different in area under the LROC curve = 0.0374, 95% CI 2-sided [0.0190 to 0.0557]

2. Secondary Outcome: The Reading Time Was Computed and Compared for Aim 1 (Baseline) and Arm 2 (With BU-CAD Assistance) Studies.
Description: Each reader's reading time of a case was automatically recorded by the BU-CAD system.
  the average reading times of 16 readers with and without outlier reading times were compared between the aided and unaided sessions using the paired t-test.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: second
Units Other Than Participants: case
Groups:
- Arm 1: Read each breast ultrasound case without the TaiHao AI assistance referred to as 'the unaided (or baseline) study
- Arm 2: Read each breast ultrasound case with the aid of BU-CAD decision support referred to as 'aided study'
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 16
Number analyzed (case) | 628 | 628
second | 31.75 [11.24 to 52.25] | 18.96 [3.25 to 34.67]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 12.78

3. Secondary Outcome: The Sensitivity, Specificity, PPV, and NPV Were Computed and Compared for Aim 1 (Baseline) and Arm 2 (With BU-CAD Assistance) Studies.
Description: The mean sensitivity, specificity, PPV, and NPV of 16 readers were calculated and compared between the aided and unaided sessions using McNemar's test.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: proportion
Units Other Than Participants: case
Groups:
- Arm 2: Read each breast ultrasound case with the TaiHao AI assistance referred to as 'the aided (or with CAD) study
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 16
Number analyzed (case) | 628 | 628
proportion
  Sensitivity | 0.9225 [0.8896 to 0.9554] | 0.9353 [0.9050 to 0.9655]
  Specificity | 0.3165 [0.2694 to 0.3636] | 0.3611 [0.3124 to 0.4098]
  PPV | 0.4876 [0.4433 to 0.5319] | 0.5056 [0.4607 to 0.5505]
  NPV | 0.8623 [0.8048 to 0.9198] | 0.8945 [0.8456 to 0.9434]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, McNemar; different in sensitivity = -0.0013, 95% CI 2-sided [-0.2307 to 0.2281]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, McNemar; different in specificity = 0.1065, 95% CI 2-sided [0.0008 to 0.2122]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, McNemar; different in PPV = -0.0860, 95% CI 2-sided [-0.1824 to 0.0104]
Statistical Analysis 4: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, McNemar; different in NPV = 0.0860, 95% CI 2-sided [-0.0104 to 0.1824]

ADVERSE EVENTS:
Time Frame: Adverse Events cannot be monitored/assessed. Because this is a retrospective reader study, not a human trial.
Description: This is a retrospective reader study. There is no adverse events and risks.
Groups:
- First Session: Manual Review First and Then Review With CADx: Each rater will interpret the "Dataset A" cases in different random order without any assistance of artificial assistance first, and then interpret the "Dataset B" cases in different random order with BR-USCAD DS.
  Reader Group X: Each rater in "Reader Group X" will interpret the "dataset A" cases in different random order without BR-USCAD DS and interpret the "dataset B" cases in different random order with BR-USCAD DS.
- First Session: Review With CADx First and Then Manual Review: Each rater will interpret the "Dataset A" cases in different random order with BR-USCAD DS first, and then interpret the "Dataset B" cases in different random order without any assistance of artificial assistance.
  Reader Group Y: Each rater in "Reader Group Y" will interpret the "dataset A" cases in different random order with BR-USCAD DS and interpret the "dataset B" cases in different random order without BR-USCAD DS.
- Second Session: Manual Review First and Then Review With CADx: At least 4 weeks after first session for memory washing out. Each rater will interpret the "Dataset A" cases in different random order without any assistance of artificial assistance first, and then interpret the "Dataset B" cases in different random order with BR-USCAD DS.
  Reader Group Y: Each rater in "Reader Group Y" will interpret the "dataset A" cases in different random order with BR-USCAD DS and interpret the "dataset B" cases in different random order without BR-USCAD DS.
- Second Session: Review With CADx First and Then Manual Review: At least 4 weeks after first session for memory washing out. Each rater will interpret the "Dataset A" cases in different random order with BR-USCAD DS first, and then interpret the "Dataset B" cases in different random order without any assistance of artificial assistance.
  Reader Group X: Each rater in "Reader Group X" will interpret the "dataset A" cases in different random order without BR-USCAD DS and interpret the "dataset B" cases in different random order with BR-USCAD DS.
Arm/Group | First Session: Manual Review First and Then Review With CADx | First Session: Review With CADx First and Then Manual Review | Second Session: Manual Review First and Then Review With CADx | Second Session: Review With CADx First and Then Manual Review
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT04551105/Prot_SAP_001.pdf